

## Statistical Analysis Plan

Protocol Version: Amendment 3

Protocol Date: November 1, 2019

Analysis Plan Version: 2.0

Analysis Plan Date: September 12, 2023

## TABLE OF CONTENTS

| 1 | I | ntro | duction | <del>(</del> |
|---|---|---|---|---|
| | 1.1 | . : | Study Design | 6 |
| | 1.2 | Stuc | dy Objectives | 6 |
| | 1 | 1.2.1 | Primary Objective | 6 |
| | 1 | 1.2.2 | Secondary Objectives | e |
| | 1.2 | : | Sample size Considerations | 7 |
| 2 | ( | Gene | eral Considerations for Data Analyses | <u>c</u> |
| | 2.1 | | Analysis Populations | <u>c</u> |
| | 2 | 2.1.1 | Intention-to-treat Population (ITT) | <u>c</u> |
| | 2 | 2.1.2 | Modified Intention-to-treat Infusion Population (mITT) | <u>c</u> |
| | 2.2 | . | Data Sources | <u>C</u> |
| | 2.3 | . ( | General Analysis Conventions | <u>c</u> |
| | 2.4 | . | Disposition of Participants | 10 |
| | 2.5 | | Demographic and Baseline Characteristics | 10 |
| | 2.6 | | Handling of Missing Data | 10 |
| 3 | A | Analy | ysis of Clinical Endpoints | 11 |
| | 3.1 | . ( | General | 11 |
| | 3 | 3.1.1 | Estimands and Censoring Scheme | 11 |
| | 3 | 3.1.2 | Event Data | 16 |
| | 3 | 3.1.3 | Assessment of Model Assumptions | 16 |
| | 3 | 3.1.4 | Multiple Comparisons and Composite Endpoints | 17 |
| | 3.2 | . | Primary Endpoint Analysis | 17 |
| | 3 | 3.2.1 | Primary Analysis | 17 |
| | 3 | 3.2.2 | Sensitivity Analyses of the Primary Outcome | 18 |
| | 3.3 | | Analysis of the Secondary Endpoints | 19 |
| | 3 | 3.3.1 | Recurrent-event analysis of the primary endpoint | 19 |
| | 3 | 3.3.2 | Time to Event Analysis of the Secondary Endpoints | 20 |
| | 3 | 3.3.3 | Sensitivity Analyses of the Secondary Outcomes | 21 |
| | 3.4 | . : | Subgroup Analyses | 21 |
| | 3.5 | . : | Safety Analyses | 22 |
| 4 | F | Refer | rences | 23 |
| 5 | ( | SAP F | Revision | 24 |

| TACT2 | Statistical | Analysis | Plan. | v 2.0: | Septemb | er 12 | 2023 |
|-------|-------------|----------|-------|--------|---------|-------|------|

#### Signature page

Electronically signed by: Hayley Nemeth Hayley Nemeth Prepared by: Reason: Approved Date: Sep 19, 2023 13:06 EDT Date Hayley Nemeth, MS **DCRI Statistics Representative** Biostatistician III **Duke Clinical Research Institute** Reviewed by: Electronically signed by: Kevin J. Anstrom Kevin J. Anstrom Reason: Approved Date: Sep 19, 2023 18:29 EDT Kevin J. Anstrom, PhD Date Co-Principal Investigator, DCC University of North Carolina Gillings School of Global Public Health Approved by: Electronically signed by: Gervasio Lamas Gervasio Lamas Reason: Approved Date: Sep 21, 2023 16:42 EDT ..... Gervasio A. Lamas, MD, Date Principal Investigator, CCC Mount Sinai Medical Center and Columbia **University Medical Center** Electronically signed by: Daniel Mark Daniel Mark Reason: Approved Date: Sep 23, 2023 18:08 EDT Daniel B. Mark, MD, MPH, Date Co-Principal Investigator, DCC **Duke Clinical Research Institute** Electronically signed by: Mario Stylianou Mario Stylianou Reason: Approved Date: Sep 25, 2023 12:07 EDT Mario Stylianou, PhD Date **NIH Representative** National Heart, Lung, and Blood Institute/National Institutes of Health

## **Abbreviations**

| Abbreviation | Definition |
|--------------|--------------------------------------------|
| CEC | Clinical Events Committee |
| CI | Confidence Interval |
| CONSORT | Consolidated Standards of Reporting Trials |
| CRF | Case Report Form |
| CSR | Clinical Study Report |
| DCRI | Duke Clinical Research Institute |
| EDC | Electronic Data Capture |
| FU | Follow-Up |
| HR | Hazard Ratio |
| ITT | Intention-To-Treat |
| MI | Myocardial Infarction |
| mITT | Modified Intention-To-Treat |
| NDI | National Death Index |
| OMVM | Oral MultiVitamins and Multiminerals |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| TACT2 | Trial to Assess Chelation Therapy 2 |
| WLW | Wei, Lin, and Weissfeld |

#### 1 Introduction

The purpose of this Statistical Analysis Plan (SAP) is to describe the analyses and data presentations that will be used for the creation of the primary manuscript of the study which will focus on the comparison of active chelation vs. placebo chelation.

#### 1.1 Study Design

The Trial to Assess Chelation Therapy 2 (TACT2) is a randomized, double blinded, placebo-controlled 2x2 factorial clinical trial. The study treatments are edetate disodium-based chelation (weekly infusion for 40 weeks) and high-dose oral multivitamins and multi-minerals (OMVM) (twice daily for up to 5 years). Subjects with diabetes mellitus with a prior myocardial infarction (MI) are recruited from participating sites in the US and Canada and randomized in a 1:1:1:1 fashion to 4 groups:

- i. Active chelation + active OMVM
- ii. Active chelation + placebo OMVM
- iii. Placebo chelation + active OMVM
- iv. Placebo chelation + placebo OMVM.

Patients will be followed for clinical events until the earlier of database lock or five years from randomization. Clinical outcomes will be collected by study sites at each infusion visit and by the DCRI Call Center at month 6 and 12, and every 4 months afterwards with the last assessment at month 60.

TACT2 is an event driven trial with a plan to continue until at least 282 primary endpoint events are identified. The original planned sample size was 1200 participants. The sample size was later modified to 1100. The final enrollment is 1000, but with an increased follow-up time to preserve statistical power. More details on sample size and power calculation are included later in the SAP.

#### 1.2 Study Objectives

TACT2 seeks to replicate TACT, which found a reduction of recurrent cardiovascular events most prominent in the subgroup of post-MI diabetic patients receiving edetate disodium-based chelation therapy.

#### 1.2.1 Primary Objective

The primary objective of TACT2 is to determine if the chelation-based strategy increases the time to the first occurrence of any of the components of the primary composite endpoint of all-cause mortality, MI, stroke, coronary revascularization, or hospitalization for unstable angina compared with the placebo chelation strategy.

#### 1.2.2 Secondary Objectives

The secondary objectives of TACT2 are to determine:

- i. if the chelation-based strategy reduces the overall rate of occurrence of the events which define the primary composite endpoint of all-cause mortality, MI, stroke, coronary revascularization, or hospitalization for unstable angina events compared with the placebo chelation strategy.
- ii. to determine if the chelation-based strategy increases the time to the first occurrence of a secondary composite endpoint of cardiovascular mortality, MI, or stroke compared with the placebo chelation strategy.
- iii. to determine if the chelation-based strategy increases the time to all-cause mortality compared with the placebo chelation strategy.

#### 1.2 Sample size Considerations

The study was originally designed to enroll 1200 participants with a minimum follow-up of 12 months. Since the enrollment was slower than projected, the DSMB conducted a blinded review of enrollment aggregate event rates, and projected event rates in July 2019. The study team proposed a new sample size based on the updated projected event rate, an assumed hazard ratio of 0.7 comparing chelation and placebo, and a dropout rate of 5% (Table 1). While the sample size was reduced to 1100 with an extended enrollment time by December 2020, the follow-up (FU) period was extended to 2 years to ensure to have the targeted power of 85%.

The final study enrollment was 1000. The study team evaluated the study power with a newly extended FU period of 2.5 years assuming various dropout rates (Table 2). Even with a dropout rate of 10%, the study power exceeds the targeted power of 85% with 1000 participants and 2.5 years of follow-up.

The full details around sample size adjustment and study power are included in Appendix I.

| Sample<br>size | Note | Power | Overall<br>event rate<br>(%/pt-yr) | Assumed<br>event rate<br>in EDTA<br>(%/pt-yr) | Assumed event rate in Placebo (%/pt-yr) | Dropout<br>rate | Enrollment<br>year | FU<br>year | Total #<br>events |
|---|---|---|---|---|---|---|---|---|---|
| 1200 | Original sample size | 85% | 10.9% | 8.97% | 12.81% | 2% | 3 | 1 | 282 |
| 1100 | Modified | 88% | 9.2% | 7.56% | 10.82% | 5% | 4.25 | 2 | 308 |

Table 1. Original and modified sample size and study power

Table 2. Study power with the final 1000 participants enrolled

| Scenario | Overall event rate (%/pt-yr) | Assumed event rate in EDTA (%/pt-yr) | Assumed event rate in Placebo (%/pt-yr) | Overall dropout rate | Mean<br>power | Mean # events |
|---|---|---|---|---|---|---|
| | | | | 5% | 89% | 299 |
| Projected | 8.8 | 7.2 | 10.4 | 7% | 88% | 295 |
| | | | | 10% | 87% | 288 |

## 2 General Considerations for Data Analyses

#### 2.1 Analysis Populations

#### 2.1.1 Intention-to-treat Population (ITT)

The ITT population will include all randomized participants, including those who are later found not to meet study eligibility criteria. There were two participants who mistakenly "re-joined" the trial after infusions ended and were re-randomized in a second site, near their original site. The detail for the two participants is in Appendix II. They will only be counted once in the ITT population. Their data from the 2<sup>nd</sup> randomization will not be included the analysis.

#### 2.1.2 Modified Intention-to-treat Infusion Population (mITT)

All participants in the ITT population who have completed at least one infusion will be included in the modified intention-to-treat population. The mITT population will be the primary analysis population.

#### 2.2 Data Sources

The data used for analysis will come from 5 sources: the randomization data from the Interactive Voice/Web System (IXRS), the e-CRF data collected by the iMedidata Rave electronic data capture system (RAVE), the adjudicated endpoint data from the clinical events committee database (CEC), the site-level information stored in the Clinical Trial Management System (CTMS) database, and the CDC National Death Index (NDI).

Masked-source NDI search results will be used to focus a search for supporting clinical and other documentation. If supporting documentation is obtained, the data will be submitted to the CEC process prior to being used in the analysis. If needed, a Mortality Review Committee will be assigned to classify potential death events when there are insufficient/incomplete or contradictory NDI and/or Call Center data to make a reliable determination. Additional details will be described in a separate charter.

#### 2.3 General Analysis Conventions

Statistical comparisons will be performed using two-sided significance tests. An alpha level of 0.05 will determine significance unless otherwise specified.

Continuous variables will be presented in terms of percentiles (e.g., median, 25th percentile, and 75th percentiles) along with means and standard deviations. Categorical variables will be summarized in terms of frequencies and percentages.

All programs written to create analysis datasets or perform analyses will be validated according to SOPs by the Statistical Programming group.

All statistical analysis will be performed using SAS® v9.4 or higher (Cary, NC USA) and/or other proper software, e. g. R.

#### 2.4 Disposition of Participants

Disposition of participants (number randomized, number who received treatment, number of infusions received per patient, number of withdrawals and dropouts from the study, number lost to follow-up, length of follow-up, time since last contact, number unmasked) will be summarized by active chelation vs placebo chelation groups using a CONSORT flow diagram and subject disposition table.

Lost to follow-up among alive and non-withdrawn participants will be reported in the CONSORT diagram as described above. The number of participants lost to follow-up with a primary endpoint will be included in the total and also reported separately. Participants alive and not withdrawn or lost to follow-up will be defined as completing the study.

The definition for lost to follow-up will be:

No contact within 12 months of the end of study. End of study is defined as the 5-year informed consent expiration date or administrative end of study date (June 30, 2023). Last contact is defined as the last known alive date.

#### 2.5 Demographic and Baseline Characteristics

Demographic and baseline characteristics will be summarized by active and placebo chelation groups and for the overall mITT population. These include cardiovascular risk factors, comorbidities, relevant descriptors from the history, concomitant medical care including post-MI medications, treatments for diabetes, over-the-counter supplements and herbal remedies. Physical examination, laboratory data, cardiopulmonary symptoms, and past clinical events. Blood and urine metals pre- and post-chelation are discussed in the SAP for the Trave Metals Biorepository Core Lab.

#### 2.6 Handling of Missing Data

Every effort will be made to obtain complete data during the course of the trial. If missing data remains despite all the efforts, rules on how to handle the missing data will be implemented.

If the proportion of subjects with missing values in any of the covariates for the primary analysis, i.e. age, sex, and baseline insulin use, is greater than 1%, then the missing values will be imputed to the mode.

Since the clinical endpoints are adjudicated by the CEC, we don't anticipate missing values for positively adjudicated outcomes. In the very rare occasion where the event day is missing, it will be imputed as the last day of the month. If missing day and month, then December 31<sup>st</sup> of the provided year will be used. If the year is missing, no imputation will be performed.

## 3 Analysis of Clinical Endpoints

#### 3.1 General

## 3.1.1 Estimands and Censoring Scheme

Summaries of the descriptions of the estimand attributes and censoring schemes are shown in **Table 3**. Like TACT, the primary analysis will include all identified events obtained as part of the planned follow-up from infusion visits and call center interviews.

Table 3. Key Study Estimands and Censoring Scheme.

| Objective Description / Study Population | Endpoint | Summary<br>statistics | Events to be included in the endpoint derivation | Censoring date |
|---|---|---|---|---|
| Primary Objective/mITT | Time from randomization to the first occurrence of primary composite endpoint of all-cause mortality, MI, stroke, coronary revascularization, or hospitalization for unstable angina | Hazard ratio estimate based on a Cox proportional hazards model. | All positively adjudicated primary endpoint events post-randomization except those occurring after withdrawal of consent or ICF expiration. Events occurring after withdrawal consent or ICF expiration will be censored. Subjects with events after withdrawal or ICF expiration will be censored at the min(date withdrew consent, date of last contact with patient/proxy where event status was assessed). | Among subjects not experiencing endpoint of interest: Censoring date = min(date withdraw consent, date of last contact with patient/proxy where event status was assessed) Date of last contact defined as: If the last contact occurred during the study infusion phase - use last infusion visit date where survival status and event status were assessed (yes or no to event). If last contact occurred during call center follow up period – use 'complete' incomplete' status date by patient/proxy where survival status and hospitalization status were assessed (yes or no to hospitalization). |

| Secondary Objective / mITT | Overall rate of recurrent events due to all-cause mortality, MI, stroke, coronary revascularization, or hospitalization for unstable angina | Hazard ratio estimate based on a proportional intensity model by Andersen-Gill and a marginal model by Wei, Lin and Weissfeld. | *same as primary endpoint | For composite endpoints, date of last assessment = the earliest of the last assessment date among all components. *same as primary endpoint |
|---|---|---|---|---|
| Secondary Objective / mITT | Time from randomization to the first occurrence of the secondary composite endpoint of cardiovascular mortality, MI, or stroke | Cause specific hazard ratio estimate based on a cause-specific Cox proportional hazards model. | All positively adjudicated endpoint events post-randomization except those occurring after withdrawal of consent or ICF expiration date. Non-CV death or undetermined cause of death is considered a competing risk. Among subjects experiencing competing risk (non-CV death or undetermined death is a competing risk of CV death or undetermined death is a competing risk of CV death or MI/stroke if a subject died without having any | Among subjects not experiencing endpoint of interest or competing event: Censoring date = min(date withdraw consent, date of last contact with patient/proxy where event status was assessed) *Date of last contact defined in 1st row, 5th column (primary endpoint) |

| | | | of these events<br>beforehand):<br>Event date = non-<br>CV or<br>undetermined<br>death date; | |
|---|---|---|---|---|
| Secondary Objective / mITT | Time from randomization to all-cause mortality | Hazard ratio estimate based on a Cox proportional hazards model. | All deaths post-randomization (including adjudicated deaths obtained from the NDI search) A death date after withdrawn consent or ICF expiration (obtained from public data source) is considered an event. | Among subjects who are alive: Censoring date = (date last known alive) Date of last known alive defined as: If the last contact occurred during the study infusion phase - use last infusion visit date. If last contact occurred during call center follow up period – use 'complete'/incomplete' status date by patient/proxy or ('not done' status date where source = patient) or last alive date from Call Center where death status was assessed. |
| Secondary Objective / mITT | Total number of SAE and percentage of patients experiencing at least 1 SAE. | Number and proportions by treatment group. Confidence intervals will be based on the Miettinen-Nurminen method. | Randomization to<br>min(withdraw<br>consent, 30 days<br>post final infusion) | N/A |

| Sensitivity Analysis of<br>the Primary Outcome<br>/ Bayesian analysis<br>using TACT results as<br>one of the priors /<br>mITT | *Same as primary<br>analysis | Treatment effect<br>mean posterior<br>hazard ratio based<br>on a Bayesian<br>time to event<br>model | *Same as primary<br>analysis | *Same as primary analysis |
|---|---|---|---|---|
| Sensitivity Analysis of<br>the Secondary All-<br>Cause Mortality<br>Outcome / Bayesian<br>analysis using TACT<br>results as one of the<br>priors / mITT | *Same as primary<br>analysis | Treatment effect<br>mean posterior<br>hazard ratio based<br>on a Bayesian<br>time to event<br>model | *Same as primary<br>analysis | *Same as primary<br>analysis |
| Sensitivity Analysis of<br>the Primary Outcome<br>/ ITT | *Same as primary analysis | *Same as primary<br>analysis | *Same as primary analysis | *Same as primary analysis |
| Sensitivity Analysis of<br>the Primary Outcome<br>/ mITT with imputed<br>event status for<br>subjects withdrew<br>/lost to follow up | *Same as primary<br>analysis | *Same as primary<br>analysis | *Same as primary analysis except that the event status will be imputed for subjects who withdrew consent or lost to follow up before study completion | *Same as primary analysis |

| Sensitivity Analysis of the Primary Outcome/ mITT with the exclusion of positively adjudicated events > 1 year after the last contact where all components of the composite were assessed | *Same as primary analysis | *Same as primary analysis | *Same as primary analysis but exclude positively adjudicated events more than 1 year from the most recent study contact where all components of the composite endpoint were assessed. | Among subjects not experiencing endpoint of interest or experiencing first CEC event > 1 year after event assessment date: Censoring date = min(date withdraw consent, date of last contact with patient/proxy where event status was assessed) *Date of last contact defined in 1st row, 5th column (primary endpoint) |
|---|---|---|---|---|
| Sensitivity Analysis of<br>the Secondary<br>Composite Outcome/<br>Where undetermined<br>death is considered<br>CV-death / mITT | *same as<br>secondary<br>composite<br>endpoint | *same as secondary composite endpoint, where: Undetermined death is analyzed as CV-death. | *same as<br>secondary<br>composite<br>endpoint | *same as secondary composite endpoint |
| Sensitivity Analysis of<br>the Secondary<br>Composite Objective /<br>Cause of death based<br>on best available data<br>(from CEC or CRF if<br>CEC is unavailable) /<br>mITT | *Same as<br>secondary<br>composite<br>analysis | *Same as<br>secondary<br>composite<br>analysis | *Same as secondary composite analysis, where: Cause of death is determined based on best available data. If cause of death from CEC is available, use CEC cause of death. Otherwise, if CRF cause of death available, use CRF cause of death. | *Same as secondary composite analysis |

| | | | If cause of death is<br>unavailable in CEC<br>and CRF, use NDI<br>cause of death. | |
|---|---|---|---|---|
| Sensitivity Analysis of<br>the Secondary All-<br>Cause Mortality<br>Outcome / Censor at<br>the date of NDI<br>assessment / mITT | *Same as<br>secondary all-<br>cause mortality<br>analysis | *Same as<br>secondary all-<br>cause mortality<br>analysis | *Same as<br>secondary all-cause<br>mortality analysis | Among subjects who are alive: Censoring date = max(date of NDI assessment, last known alive date) Date of NDI assessment is defined as: The last date that NDI results were assessed. This will be consistent for all participants without an event. |

<sup>\*</sup>See section 2.1 for the definition of ITT and mITT.

One participant who was randomized twice and received infusions from the second site will be censored at the second randomization. The other participant who was lost to follow-up at the first site and then was randomized at the second site will be censored at the time of lost to follow-up at the first site.

#### 3.1.2 Event Data

Analyses of the clinical endpoints will use the CEC-adjudicated data for death, MI, stroke, coronary revascularization, or hospitalization for unstable angina.

#### 3.1.3 Assessment of Model Assumptions

The validity of the proportional hazards assumption will be examined using a standard graphical method such as Schoenfeld residual plots. If the assumption holds, the survival curves should be approximately parallel to each other. An additional analytical method that includes the supremum test as implemented by using the ASSESS statement in PROC PHREG in SAS version 9.4 may be utilized. A *P*-value of < 0.05 indicates violation of the proportional hazards assumption. If there is evidence of non-proportionality, a time dependent covariate will be included in the model, or a restricted mean survival time model will be performed.

#### 3.1.4 Multiple Comparisons and Composite Endpoints

With the number of primary hypotheses and the various secondary endpoints to be analyzed and compared, there is an increased probability that at least one of the comparisons could be "significant" by chance. We have pre-specified the primary and secondary outcome variables to help avoid over-interpretation and to reduce the problems inherent with multiple testing. We will be conservative in the interpretation of these analyses, taking into account the degree of significance, and looking for consistency across endpoints.

#### 3.2 Primary Endpoint Analysis

The primary endpoint is the composite of all-cause mortality, MI, stroke, coronary revascularization, or hospitalization for unstable angina.

If two of the component events of the primary composite endpoint occur on the same day, the following hierarchy will be used when reporting the components of the primary endpoint. For example, a patient with stroke and all-cause mortality on the same date will be considered as having stroke when summarizing individual events within the primary composite outcome. This hierarchy will only be used for summarizing events within the primary composite outcome and will not affect the primary analysis.

- i. MI
- ii. Stroke
- iii. Hospitalization for unstable angina
- iv. Coronary revascularization
- v. All-cause mortality

#### 3.2.1 Primary Analysis

The primary objective is to determine if the chelation-based strategy increases the time to composite endpoint compared with the placebo chelation strategy. The primary composite endpoint will be analyzed using a Cox proportional hazards regression model of time from randomization to the first occurrence of all-cause mortality, MI, stroke, coronary revascularization, or hospitalization for unstable angina.

The primary analysis will be based on a Cox model which includes indicator variables for the active chelation as the primary variable of interest and active OMVM groups, age, sex, and baseline insulin use as covariates. Age will be included in the model in the form of cubic splines using three knots at 10<sup>th</sup>, 50<sup>th</sup>, and 90<sup>th</sup> percentiles. Two separate manuscripts will explore the effect of active OMVM and the effects of chelation by OMVM.

The chelation treatment effect will be summarized using hazard ratios and associated 95% Cls. A hazard ratio of < 1 would suggest a benefit for the chelation-based therapy. Kaplan Meier survival estimates will be constructed based on the time from randomization to the first

primary event occurrence. Events occurring after withdrawal of consent or informed consent expiration will be censored.

The OMVM treatment effect from the Cox model will be estimated using the Cox model described above. A hazard ratio of < 1 would suggest a benefit for OMVM treatment. Given the focus on chelation therapy, the interpretation of the OMVM treatment effect will be considered exploratory. A full set of analyses of the 2x2 design will be reported in a separate manuscript.

Four interim analyses were conducted at 25%, 40%, 60%, and 80% of expected information using a Haybittle-Peto-type boundary for efficacy (i.e. p<=0.001, Z=3). For this reason, the adjusted two-sided significance level for the final analysis is 0.05 (i.e., the corresponding critical value, Z = -1.96).

Formal statistical hypothesis testing will follow a hierarchy based on statistical significance of the prior endpoint. If the prior endpoint is statistically significant at the 0.05 level, the next endpoint's p-value will be tested for significance. The outcome hierarchy will be evaluated as follows:

- 1) Primary composite outcome
- 2) Secondary all-cause mortality outcome (with conservative censoring)
- 3) Secondary composite outcome of cardiovascular mortality, MI, or stroke
- 4) Secondary recurrent event analysis (Andersen & Gill method)

#### 3.2.2 Sensitivity Analyses of the Primary Outcome

The primary hypothesis for the primary composite endpoint will be tested using the ITT population as a sensitivity analysis.

A sensitivity analysis was initially planned to investigate the potential effect of the COVID-19 outbreak on the primary analysis. Instead, the potential effect of COVID-19 may be explored in a separate manuscript.

A sensitivity analysis will use Bayesian methods to estimate the primary outcome treatment effect posterior distribution using the first TACT trial results and other related information to develop a set of priors for the treatment effect (Zampieri, 2020). As suggested by Zampieri, these analyses will include at least one prior distribution for the effect of chelation vs. placebo in each of the following categories: skeptical, pessimistic, and optimistic. The priors will be assumed to follow a normal distribution and will represent the log hazard ratio from the Cox model. There will be two skeptical (non-informative) priors for the log hazard ratio with a mean of zero and differing standard deviations (e.g., one standard deviation will be 10 and the other will be 100). Two pessimistic priors for the log hazard ratio will also be included, both will be centered around zero and allow for low probability of a favorable treatment effect (e.g., 0.5%

and 2.5% probability of the hazard ratio for chelation of 0.80 compared to placebo). The two optimistic priors will include the overall treatment effect from TACT (e.g., HR of 0.82 with a 95% CI of 0.69 to 0.99) and diabetes subgroup treatment effect from TACT (e.g., HR of 0.59 with a 95% CI of 0.44 to 0.79). In all of the above models, the priors for the parameters associated with other model covariates will be non-informative with large standard deviations (e.g., standard deviation of 100) and center at zero for the associated log hazard ratios. The chelation treatment effect will be summarized using mean posterior hazard ratios and associated 95% highest posterior density credible intervals. A mean posterior hazard ratio of < 1 would suggest a benefit for the chelation-based therapy.

Another sensitivity analysis is planned to assess how the primary analysis would be affected by various assumptions regarding the occurrence of primary endpoint events among those who withdrew consent or were lost to follow-up, as was performed and published in TACT. Baseline characteristics by treatment group will be assessed for the patients who did versus did not withdraw consent or were lost to follow-up. Events will be imputed by simulation only for the consent withdrawal or lost patients who did not have a documented occurrence of one of the primary events prior to the withdrawn consent/lost to follow-up. The different percentages of the withdrawn or lost patients will be assumed to have an event at their censoring time. The event rates among patients that withdrew or were lost to follow-up in each treatment group will be varied across a broad spectrum and include scenarios that were markedly unfavorable to chelation. The imputed event rates for patients who withdrew consent or were lost to follow-up will be combined with the observed event rates of patients who completed the study to assess the treatment effect via a hazard ratio. These analyses will focus on scenarios in which events among withdrawn or lost patients in the active arm are assumed to occur at a higher rate than withdrawn or lost patients in the placebo arm.

Another sensitivity analysis is planned for the primary endpoint to censor, at the point of last contact, those deaths that were identified more than one year following the most recent study contact.

#### 3.3 Analysis of the Secondary Endpoints

The three secondary endpoints are:

- i. Recurrent events of the primary composite endpoint
- ii. All-cause mortality
- iii. Composite of cardiovascular mortality, MI, or stroke

#### 3.3.1 Recurrent-event analysis of the primary endpoint

Recurrent event analyses include all positively adjudicated primary endpoint events attributed to a participant: all-cause mortality, recurrent MI, stroke, coronary revascularization, or hospitalization for unstable angina events. The number of patients with a primary composite endpoint and the frequency of the primary composite endpoint per each component will be

summarized by active chelation and placebo. We analyze this endpoint using two statistical techniques:

- i. The generalization of the Cox model to handle recurrent events developed by Andersen & Gill (1982) is the most frequently used approach to estimate treatment differences with total and recurrent events. This approach models gap time (time from enrollment to first event or from one event to the next) and assumes independence of observed event times within the same subject with the adjustment of the covariates. Our modeling will use robust standard errors to account for individual patients' heterogeneity and covariance across event times. The treatment effect will be presented as a hazard ratio (EDTA vs. placebo) and associated 95% CIs and *P*-value. It will be the primary analysis for the total number of all-cause mortality, recurrent MI, stroke, coronary revascularization, or hospitalization for unstable angina events endpoint.
- ii. The stratified marginal Cox modeling approach developed by Wei, Lin, and Weissfeld (WLW) (1989) considers each event recurrence separately and models all the available data for the specific event. Therefore, each subject is considered to be at risk for all events, regardless of how many events each subject actually experienced. A different baseline hazard function is assumed for each event, through use of strata for each event. The WLW will model the marginal hazard of each event's failure time. The time interval for each event for each subject starts at date of randomization and ends at the time of the specific event or censoring. A treatment effect will be presented as a hazard ratio (EDTA vs. placebo) and a 95% CI and *P*-value. This will be considered as a sensitivity analysis.

Both analyses will be adjusted for age, sex, and baseline insulin use. In either analysis, a hazard ratio of < 1 would suggest a benefit for the chelation-based therapy.

An event rate of the endpoint for each treatment group will be calculated as percentage per 100 patient years, accounting for differential follow-up duration. A 95% CI for the event rates will be calculated as

$$(\frac{r_C}{T_C}) \pm 1.96\sqrt{\frac{r_C}{T_C^2}},$$

where subscript C denotes the chelation arm, and r is the total number of event occurrences, and T is the total follow-up time among all participants.

#### 3.3.2 Time to Event Analysis of the Secondary Endpoints

The analyses for the time to the first occurrence of secondary endpoints (1) time to the first occurrence of the composite of cardiovascular mortality, MI, or stroke; 2) time to all-cause

mortality) will be performed in the same manner as the primary analysis in Section 4.1, replacing the primary composite endpoint with secondary endpoints.

Competing risk of non-CV death or undetermined death will be taken into account for the secondary composite endpoint (time to the first occurrence of the composite of cardiovascular mortality, MI, or stroke). Follow-up will be censored at the time of non-CV or undetermined death if there is no prior composite event. For this endpoint, the treatment effect will be presented as a cause-specific hazard ratio.

All deaths post-randomization will be included in the secondary all-cause mortality endpoint. For this endpoint, a death date after withdrawal of consent or ICF expiration (obtained from public data sources) is considered an event.

#### 3.3.3 Sensitivity Analyses of the Secondary Outcomes

A sensitivity analysis is planned for the secondary composite endpoint where undetermined death will be classified as CV-death.

Another sensitivity analysis is planned for the secondary composite endpoint where cause of death is determined based on the best available data. Cause of death will first be determined based on the data from the CEC. If cause of death from the CEC is unavailable, cause of death will be determined from the CRF data. If cause of death from the CEC and CRF is unavailable, cause of death will be determined based on the NDI data.

A sensitivity analysis is planned for the secondary all-cause mortality endpoint where participants with no event will be censored at the last date that NDI results were assessed. The censoring date will be consistent for all participants without an event.

A sensitivity analysis will use Bayesian methods to estimate the secondary all-cause mortality outcome treatment effect posterior distribution. These analyses will be performed in an analogous manner as the Bayesian analysis of the primary outcome (section 3.2.2).

#### 3.4 Subgroup Analyses

To examine the heterogeneity of the treatment effect, subgroup analyses for the primary and secondary endpoints will be performed using interaction terms within the Cox proportional hazards model. The pre-specified key subgroups of interest are following.

- Sex: female vs. male
- Race: White vs. Black vs. Other
- Ethnicity: Hispanic vs. non-Hispanic (unknown ethnicity is considered missing)
- Age: ≤ 70 years vs. > 70 years
- MI location: anterior MI vs. non-anterior MI

- Pharmacologic treatment of diabetes (two subgroups analyses: no insulin vs. insulin, SGLT2i or GLP-1a vs. neither)
- Known peripheral artery disease at baseline: yes vs. no
- Tertiles of lead (in blood) and cadmium (in urine)

For categorical variables, if the proportional hazards assumption is violated, we will include the subgroup factor as a stratification variable within the Cox regression model. This model structure will decrease the reliance on the proportional hazards assumption. Event rates by treatment and HRs with 95% CIs will be reported for each subgroup. Forest plots will be generated displaying the estimated hazard ratios and 95% CIs for each subgroup. For subgroups defined using continuous variables, the analysis based on the continuous form will be considered primary but for display purposes these variables can also be categorized.

To further analyze the heterogeneity of treatment effects at the patient level, a separate manuscript will use the PATH statement approach for subgroup analyses.

The use of statin treatment at baseline will be evaluated as a subgroup analysis in the OMVM manuscript.

#### 3.5 Safety Analyses

Using the mITT population, the total number of serious adverse events (SAEs) and percentage of participants experiencing at least one SAE from randomization to 30 days post final infusion in each patient group will be compared with confidence intervals based on the Miettinen-Nurminen method. Whether SAEs were associated with treatment and required hospitalization (inpatient hospitalization or prolongation of existing hospitalization) will be summarized per Body System or Organ Class and Dictionary-Driven Term.

#### 4 References

Andersen, P. K., & Gill, R. D. (1982). Cox's regression model for counting processes: a large sample study. *The Annals of Statistics*, 1100-1120.

Finkelstein, D. M., & Schoenfeld, D. A. (1999). Combining mortality and longitudinal measures in clinical trials. *Statistics in Medicine*, 18(11), 1341-1354.

Lamas GA, Anstrom KJ, Navas-Acien A, Boineau R, Kim H, Rosenberg Y, Stylianou M, Jones TLZ, Joubert BR, Santella RM, Escolar E, Aude YW, Fonseca V, Elliott T, Lewis EF, Farkouh ME, Nathan DM, Mon AC, Gosnell L, Newman JD, Mark DB; TACT2 Investigators. The trial to assess chelation therapy 2 (TACT2): Rationale and design. *Am Heart J.* 2022 Oct;252:1-11. doi: 10.1016/j.ahj.2022.05.013. Epub 2022 May 19. PMID: 35598636.

Lamas GA, Goertz C, Boineau R, Mark DB, Rozema T, Nahin RL, Drisko JA, Lee KL. Design of the Trial to Assess Chelation Therapy (TACT). *Am Heart J.* 2012 Jan;163(1):7-12. doi: 10.1016/j.ahj.2011.10.002.

Luo, X., Tian, H., Mohanty, S., & Tsai, W. Y. (2015). An alternative approach to confidence interval estimation for the win ratio statistic. *Biometrics*, 71(1), 139-145.

TACT Final Study SAP. (NCT00044213) https://classic.clinicaltrials.gov/ct2/show/NCT00044213

https://biolincc.nhlbi.nih.gov/studies/tact/#:~:text=Design,regimen%20or%20an%20oral%20pl acebo.

Wei, L. J., Lin, D. Y., & Weissfeld, L. (1989). Regression analysis of multivariate incomplete failure time data by modeling marginal distributions. *Journal of the American Statistical Association*, 84(408), 1065-1073.

Zampieri FG, Casey JD, Shankar-Hari M; Harrell Jr. FE, and Harhay MO (2021). "Using Bayesian Methods to Augment the Interpretation of Critical Care Trials: An Overview of Theory and Example Reanalysis of the Alveolar Recruitment Trial." *Am J Respir Crit Care Med*; 203(5): 543-552.

## 5 SAP Revision

| Revision Date<br>MMM dd, yyyy | Section | Summary of Revision | Reason for Revision |
|---|---|---|---|
| SEP 12, 2023 | 2.2 Data sources, 2.6 Missing data, 3.1.1 Estimands and censoring, 3.2.1 Primary Analysis, 3.2.2, Sensitivity, 3.3.1 Recurrent events, 3.4 Subgroup analyses, Appendix III | Added NDI as a data source. Updated imputation for missing data. Added sensitivity analyses. Added hierarchy for formal hypothesis testing. Added event rate equation for recurrent event analysis. Updated subgroup analyses. Added Bayesian sensitivity analysis. | Additional information on NDI. Missing dates in the data. Additional sensitivity analyses requested. Requests from PIs. |

## 6 Appendices

### Appendix I. TACT2 Sample size and study power projections as of March 1, 2021

#### 1. Enrollment and timeline

a. 1000 patients enrolled.

| Last rand subject infusion | Last rand subject Follow-up | Last endpoint adjudicated | Database lock |
|---|---|---|---|
| December 2021 | June 2023 | August 2023 | October 2023 |

#### 2. Event rate in the TACT diabetic cohort (n=633)

a. EDTA: 7.8%/pt-yr = 80 events / 1031 patient-years

b. Placebo: 13.2%/pt-yr = 117 events / 886 patient-years

c. Hazard ratio: 0.59

#### 3. Original and modified sample size and power

| | | | | | | | Assumed | |
|---|---|---|---|---|---|---|---|---|
| | | | | | Overall | Assumed | event | |
| | | | | | event | event | rate | |
| | | | | | rate | rate | in | |
| Sample | | | | Hazard ratio | (%/pt- | in EDTA | Placebo | Total # |
| size | Enrollment | FU | Power | (EDTA/placebo) | yr) | (%/pt-yr) | (%/pt-yr) | events |
| 1200 | 3 years | 1<br>year | 85% | 0.7 | 10.9 | 8.97 | 12.81 | 282 |
| 1100 | 3 years +<br>15 months | 2<br>years | 88% | 0.7 | 9.2 | 7.56 | 10.82 | 308 |

#### 4. Statistical power with 1000 enrolled participants as of March 1, 2021

- As of February 23, 2021, 137 patients with at least one adjudicated primary endpoint,
   1990 patient-years from 1000 enrolled patients
  - i. Proportion of reported events adjudicated as primary endpoints = 69%
  - ii. Projected overall event rate: If 39 patients had an adjudicated primary endpoint out of 57 additional patients with at least one reported event, 176/1990 = 8.8%/pt-yr
  - iii. Minimum overall event rate: 137/1990 = 6.9%/pt-yr
  - iv. Optimistic overall event rate: If 45 patients had an adjudicated primary endpoint out of 57 additional patients with at least one reported event, 182/1990 = 9.1%/pt-yr
- b. Assumptions for simulations with 10K iterations per scenario
  - i. No re-consent for those who run out 5 years from the initial consent
  - ii. Constant parameters: a two-sided alpha=0.05, hazard ratio of EDTA to placebo=0.7, sample size=1000, FU=2.5 years
  - iii. Overall dropout rate: 5, 7, 10%
  - iv. Overall event rate: 6.9, 8.8, 9.1%/pt-yr

| Scenario | Overall<br>event rate<br>(%/pt-yr) | Assumed event rate in EDTA (%/pt-yr) | Assumed event rate in Placebo (%/pt-yr) | Overall<br>dropout rate | Mean<br>power | Mean #<br>events |
|---|---|---|---|---|---|---|
| | | | | 5% | 89% | 299 |
| Projected | 8.8 | 7.2 | 10.4 | 7% | 88% | 295 |
| | | | | 10% | 87% | 288 |
| | | | | 5% | 78% | 244 |
| Minimum | 6.9 | 5.7 | 8.1 | 7% | 77% | 240 |
| | | | | 10% | 76% | 235 |
| | | | | 5% | 88% | 307 |
| Optimistic | 9.1 | 7.5 | 10.7 | 7% | 87% | 303 |
| | | | | 10% | 86% | 297 |

#### Appendix II. Details of two participants who were randomized from two different sites

#### **Double randomization case 1**

One participant was randomized again in a neighboring site right after completing 40 infusions from the first site where randomized for the first time. The study team found out the second randomization after the participant finished 35 infusions at the second site. This participant has been actively followed up by the Call Center. This participant will be censored at the time of the second randomization for any analyses using the ITT or mITT populations.

#### **Double randomization case 2**

The other participant was lost to follow up after the third infusion at the first site and then randomized again in a neighboring site after a break of longer than a year. The participant did not receive any infusion from the second site. The Call Center was not able to locate the participant for any follow-up calls. This participant will be censored at the time of lost to follow-up at the first site for any analyses using the ITT or mITT populations.

## Appendix III. TACT2 Statistical Team

| Team | Name | Email | Attends DSMB<br>Meetings |
|---|---|---|---|
| Blinded Statistical<br>Team | Hayley Nemeth | Hayley.nemeth@duke.edu | Х |
| | Jun Wen | Jun.Wen@duke.edu | X |
| | Zhen Huang | zhen.huang@duke.edu | Х |
| | Hwasoon Kim | hwasoon.kim@duke.edu | X (left DCRI in June,<br>2022) |
| | Kevin Anstrom | kevin.anstrom@unc.edu | Х |
| Unblinded<br>Statistical Team | Yuliya Lokhnygina | yuliya.lokhnygina@duke.edu | Х |
| | Dianne Gallup | dianne.gallup@duke.edu | Х |
| | Peter Merrill | Peter.merrill@duke.edu | X (left DCRI in October,<br>2022 |
| Metals Manuscript | Zhen Huang | zhen.huang@duke.edu | Х |
| | Steve McNulty | steven.mcnulty@duke.edu | |
| | Peter Merrill | Peter.merrill@duke.edu | X (left DCRI in October, 2022) |
| | Yuliya Lokhnygina | yuliya.lokhnygina@duke.edu | X |
| NHLBI<br>Biostatistician | Mario Stylianou | stylianm@nhlbi.nih.gov | Х |
| TACT2 Project<br>Leaders | Shelby Morgan | Shelby.morgan@duke.edu | Х |
| | Anne-Marie Elliott | Ann.elliott@duke.edu | X |
| | Ana Mon | Ana.Mon@msmc.com | X |
| | Leigh Gosnell | Leigh.gosnell@duke.edu | X (Prior Project Leader) |
| | Wanda Parker | Wanda.parker@duke.edu | X (Prior Project Leader) |

# TACT2\_SAP\_primary\_manuscript\_V2.0\_2023\_0 9 12

Final Audit Report 2023-09-25

Created: 2023-09-19

By: Hayley Nemeth (hn58@duke.edu)

Status: Signed

Transaction ID: CBJCHBCAABAAAUNiGrumb3uY8zl\_vHj6RCHwHfRwUk39

# "TACT2\_SAP\_primary\_manuscript\_V2.0\_2023\_09\_12" History

- Document created by Hayley Nemeth (hn58@duke.edu) 2023-09-19 5:03:57 PM GMT- IP address: 136.226.51.16
- Document emailed to hayley.nemeth@duke.edu for signature 2023-09-19 5:05:19 PM GMT
- Email viewed by hayley.nemeth@duke.edu 2023-09-19 5:05:45 PM GMT- IP address: 136.226.51.16
- Signer hayley.nemeth@duke.edu entered name at signing as Hayley Nemeth 2023-09-19 5:06:03 PM GMT- IP address: 136.226.51.16
- Document e-signed by Hayley Nemeth (hayley.nemeth@duke.edu)

Signing reason: Approved

Signature Date: 2023-09-19 - 5:06:05 PM GMT - Time Source: server- IP address: 136.226.51.16

- Document emailed to kevin.anstrom@unc.edu for signature 2023-09-19 5:06:07 PM GMT
- Email viewed by kevin.anstrom@unc.edu 2023-09-19 - 10:28:55 PM GMT- IP address: 152.2.57.199
- Signer kevin.anstrom@unc.edu entered name at signing as Kevin J. Anstrom 2023-09-19 10:29:14 PM GMT- IP address: 152.2.57.199

Signing reason: Approved

Signature Date: 2023-09-19 - 10:29:16 PM GMT - Time Source: server- IP address: 152.2.57.199

Document emailed to gervasio.lamas@msmc.com for signature 2023-09-19 - 10:29:19 PM GMT



Email viewed by gervasio.lamas@msmc.com 2023-09-21 - 8:41:28 PM GMT- IP address: 198.179.5.251

Signer gervasio.lamas@msmc.com entered name at signing as Gervasio Lamas 2023-09-21 - 8:42:23 PM GMT- IP address: 198.179.5.251

Document e-signed by Gervasio Lamas (gervasio.lamas@msmc.com)

Signing reason: Approved

Signature Date: 2023-09-21 - 8:42:25 PM GMT - Time Source: server- IP address: 198.179.5.251

Document emailed to daniel.mark@duke.edu for signature 2023-09-21 - 8:42:27 PM GMT

Email viewed by daniel.mark@duke.edu 2023-09-21 - 8:45:46 PM GMT- IP address: 104.28.39.144

Email viewed by daniel.mark@duke.edu 2023-09-22 - 10:10:29 PM GMT- IP address: 76.182.14.163

Email viewed by daniel.mark@duke.edu 2023-09-23 - 10:03:56 PM GMT- IP address: 76.182.14.163

Signer daniel.mark@duke.edu entered name at signing as Daniel Mark 2023-09-23 - 10:08:11 PM GMT- IP address: 76.182.14.163

Document e-signed by Daniel Mark (daniel.mark@duke.edu)

Signing reason: Approved

Signature Date: 2023-09-23 - 10:08:13 PM GMT - Time Source: server- IP address: 76.182.14.163

Document emailed to stylianm@nhlbi.nih.gov for signature 2023-09-23 - 10:08:14 PM GMT

Email viewed by stylianm@nhlbi.nih.gov
2023-09-23 - 10:18:51 PM GMT- IP address: 128.231.125.178

Email viewed by stylianm@nhlbi.nih.gov 2023-09-25 - 3:44:35 AM GMT- IP address: 172.226.66.107

Signer stylianm@nhlbi.nih.gov entered name at signing as Mario Stylianou 2023-09-25 - 4:07:23 PM GMT- IP address: 108.51.245.87

Document e-signed by Mario Stylianou (stylianm@nhlbi.nih.gov)

Signing reason: Approved

Signature Date: 2023-09-25 - 4:07:25 PM GMT - Time Source: server- IP address: 108.51.245.87

Agreement completed.

2023-09-25 - 4:07:25 PM GMT

